CLINICAL TRIAL: NCT01036854
Title: Parallel, Group, Laboratory-Blinded, Single and Multiple-dose Pharmacokinetic Study of Ondansetron Administered as the Immediate-Release (Zofran) and Modified-Release (EUR1025) Formulations
Brief Title: Pharmacokinetic Study of Ondansetron Administered as IR (Zofran) and MR (EUR1025)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ODO-P8-690
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Nausea
Keywords: Ondansetron, EUR-1025
MeSH Terms: conditions — Nausea | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Regime 1 (Experimental): Regime 1 will be orally administered once daily in the morning over 6 consecutive days.
  Interventions: Drug: EUR-1025
- Regime 2 (Active Comparator): Regime 2 will be orally administered twice daily at 12 hours interval (morning and evening) over 6 consecutive days
  Interventions: Drug: EUR-1025
- Regime 3 (Active Comparator): Regime 3 will be orally administered three times daily at 8 hour intervals (morning, afternoon, evening) over 6 consecutive days.
  Interventions: Drug: EUR-1025
- Regime 4 (Experimental): Regime 4- Day 1- a single dose will be given. Day 2- one placebo capsule; Day 3- a single dose will be given . Day 4 & 5- two placebo capsules on each day; Day 6- a single does will be given.
  Interventions: Drug: EUR-1025

INTERVENTIONS:
Drug: EUR-1025 — orally, 24 mg, daily for 6 days
  Other Names: Ondansetron
  Arms: Regime 1
Drug: EUR-1025 — orally, 8 mg, twice daily over 6 consecutive days
  Other Names: Ondansetron
  Arms: Regime 2
Drug: EUR-1025 — orally, 8 mg, three times a day over 6 consecutive days
  Other Names: Ondansetron
  Arms: Regime 3
Drug: EUR-1025 — orally, 8 mg, 16 mg, 24 mg, daily, for 6 days
  Other Names: Ondansetron
  Arms: Regime 4

SUMMARY:
The objective of the study is to assess blood levels of ondansetron (EUR1025 24 mg) dose and Zofran 8 mg dose after single and multiple doses are given when taken with a meal and taken on an empty stomach.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the pharmacokinetics (PK) of ondansetron administered as a novel modified-release formulation (EUR1025 24 mg) as well as the immediate-release formulation (Zofran 8 mg) after single and multiple oral dose administration under fasting and fed conditions based on the requirements of the respective indications. The safety profile of each treatment will also be assessed by recording the nature, severity, frequency, duration and relation to the treatment of any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers
* Non- or ex-smokers
* At least 21 years of age but not older than 55 years
* Body mass index targeted to be at least 18.5 and less than 30 kg/m2.
* Acceptable lab tests
* Normal 12 lead ECG
* Negative human chorionic gonadotropin (hCG) for females.

Exclusion Criteria:

* No known hypersensitivity to Ondansetron or any related products
* No presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption
* No presence of significant heart disease or disorder discovered on screening ECG
* Not pregnant
* No alcohol or drug abuse history
* No use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP)
* No previous Investigational Product (in another clinical trial) or donated 50 ml or more of blood in the previous 28 days before day 1 of this study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Ondansetron plasma concentrations will be measured by using a validated HPLC/MS assay. | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, M.D., Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma INc., Mount Royal, Quebec, Canada